CLINICAL TRIAL: NCT00212992
Title: A Pilot Randomized Controlled Trial to Compare Fixed Versus Escalating Energy Regimens for Biphasic Waveform Defibrillation
Brief Title: Biphasic Defibrillation Study: Trial to Compare Fixed Versus Escalating Energy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2001266-01H
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest
Keywords: defibrillation; ventricular fibrillation; heart arrest
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed lower-energy (Active Comparator): Out-of-hospital cardiac arrest patients undergoing defibrillation received a fixed lower-energy regimen of 150 J for all shocks
  Interventions: Procedure: Fixed lower-energy defibrillation
- Escalating higher-Energy (Active Comparator): Out-of-hospital cardiac arrest patients undergoing defibrillation received an escalating higher-energy regimen beginning with 200 J, proceeding to 300 J for the second shock and 360 J for all remaining shocks
  Interventions: Procedure: Escalating higher-energy defibrillation

INTERVENTIONS:
Procedure: Fixed lower-energy defibrillation — Every shock administered at 150 J
  Arms: Fixed lower-energy
Procedure: Escalating higher-energy defibrillation — First shock administered at 200 J, second shock at 300 J, all subsequent shocks at 360 J
  Arms: Escalating higher-Energy

SUMMARY:
This study will compare the effect of constant low-level energy [150 joules] to an escalating energy [200-300-360 joules] regimen of biphasic waveform defibrillation on multiple patient outcomes.

DETAILED DESCRIPTION:
This pilot, which will enroll 200 subjects, will allow a reasonable estimate of effect size and this will, in turn, allow for the accurate design and planning of a definitive randomized controlled trial. The following outcomes will be evaluated:

1. Important Clinical Outcomes:

   * Successful conversion,
   * Resuscitation to one hour,
   * Survival to hospital discharge,
   * Neurological function, and
   * Quality of life.
2. Process Outcomes:

   * Number of shocks required,
   * Recurrences of VF, and
   * Responsiveness to varying periods of pulselessness.
3. Adverse Outcomes:

   * Myocardial damage.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed cardiac arrest out-of-hospital requiring defibrillation and given by first responder using an automated external defibrillator

Exclusion Criteria:

* Terminal illness or do-not-resuscitate (DNR) status
* No cardiopulmonary resuscitation (CPR) x 10 minutes
* Acute trauma
* Exsanguination
* Cardiac arrest experienced while in hospital

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2001-03 (Actual); Primary Completion 2005-09 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stiell, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stiell IG, Walker RG, Nesbitt LP, Chapman FW, Cousineau D, Christenson J, Bradford P, Sookram S, Berringer R, Lank P, Wells GA. BIPHASIC Trial: a randomized comparison of fixed lower versus escalating higher energy levels for defibrillation in out-of-hospital cardiac arrest. Circulation. 2007 Mar 27;115(12):1511-7. doi: 10.1161/CIRCULATIONAHA.106.648204. Epub 2007 Mar 12. PMID 17353443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Started | 114 | 107
Completed | 114 | 107
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Lower-energy | Escalating Higher-energy | Total
Number analyzed (Participants) | 114 | 107 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (14.2) | 66.1 (14.5) | 66.0 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 44
  Male | 88 | 89 | 177
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 114 | 107 | 221
Initial Rhythm [Count of Participants; unit: Participants]
  VT/VF | 103 | 103 | 206
  Asystole | 6 | 0 | 6
  Pulseless electrical activity | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Successful Conversion to an Organized Heart Rhythm
Time Frame: Termination of defibrillation
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Number analyzed (Participants) | 114 | 107
Participants | 28 | 39

2. Secondary Outcome: Survival to Hospital Discharge
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Number analyzed (Participants) | 114 | 107
Participants | 19 | 17

3. Secondary Outcome: Resuscitation for Survival to One Hour
Time Frame: One hour from termination of defibrillation
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Number analyzed (Participants) | 114 | 107
Participants | 54 | 44

4. Secondary Outcome: Neurologic Function
Description: The Cerebral Performance Category Score (CPC) is a five-point scale used to assess neurological outcomes after cardiac arrest. The best score, 1, indicates good cerebral performance. The worst score, 5, represents brain death.
Time Frame: 30 days
Population: Patients who survived to hospital discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Number analyzed (Participants) | 19 | 17
score on a scale | 2 [1 to 3] | 2 [1 to 2]

5. Secondary Outcome: Return of Spontaneous Circulation
Time Frame: Termination of defibrillation
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Number analyzed (Participants) | 114 | 107
Participants | 58 | 52

6. Secondary Outcome: Survival to 24 Hours
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Number analyzed (Participants) | 114 | 107
Participants | 37 | 38

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Fixed Lower-energy | Escalating Higher-energy
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/107
Other Adverse Events (participants affected / at risk) | 0/114 | 0/107

LIMITATIONS AND CAVEATS:
None applicable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No